CLINICAL TRIAL: NCT03010501
Title: Effect of Energy Density Over 5 Days in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ChildFood502; R01DK082580 (NIH)
Record Dates: First submitted 2016-12-22; First posted 2017-01-05 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100% Food Energy Density (Experimental): Baseline Food Energy Density
  Interventions: Other: Food Energy Density
- 80% Food Energy Density (Experimental): Lower Food Energy Density
  Interventions: Other: Food Energy Density
- 120% Food Energy Density (Experimental): Higher Food Energy Density
  Interventions: Other: Food Energy Density

INTERVENTIONS:
Other: Food Energy Density — Food Energy density manipulated

SUMMARY:
In this study, the investigators will vary the energy density of foods served during three 5-day periods. There will be a baseline condition, and then a condition where the energy density of food is lower and a condition where the energy density of food is higher. The primary aim is to determine the effect of varying the energy density of foods served over 5 days on energy intake in preschool children. It is hypothesized that mean daily energy intake will be greater when children are served higher energy dense foods over 5 days than when served lower energy dense foods over the same period. Additionally, it is hypothesized that daily energy intake in the conditions with higher and lower energy densities will begin to converge across the 5-day period.

ELIGIBILITY:
Inclusion Criteria:

* Attending one of the designated daycare centers

Exclusion Criteria:

* Food Allergies
* Food restrictions
* Health Issues that Preclude Participation
* Not available for duration of the study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Rolls, Principal Investigator — Penn State University
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Rolls BJ, Roe LS, Keller KL. Children's Energy Intake Generally Increases in Response to the Energy Density of Meals but Varies with the Amounts and Types of Foods Served. Am J Clin Nutr. 2024 Jan;119(1):185-195. doi: 10.1016/j.ajcnut.2023.10.019. Epub 2023 Oct 27. PMID 37890673
- [Derived] Roe LS, Keller KL, Rolls BJ. Food Properties and Individual Characteristics Influence Children's Intake Across Multiple Days of Weighed Assessments in Childcare Programs. J Nutr. 2023 May;153(5):1646-1655. doi: 10.1016/j.tjnut.2023.03.025. Epub 2023 Mar 24. PMID 36965692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children aged 3 to 5 years old were recruited from classrooms at three childcare centers in State College, PA by distributing letters to parents between September 2016 and September 2017.
Groups:
- 80% Food Energy Density First, Then 100%, Then 120%: Participants in the classroom that received the three food energy density interventions across the three periods in the order of 80%, then 100%, then 120%.
- 100% Food Energy Density First, Then 120%, Then 80%: Participants in the classroom that received the three food energy density interventions across the three periods in the order of 100%, then 120%, then 80%.
- 120% Food Energy Density First, Then 80%, Then 100%: Participants in the classroom that received the three food energy density interventions across the three periods in the order of 120%, then 80%, then 100%.
- 80% Food Energy Density First, Then 120%, Then 100%: Participants in the classroom that received the three food energy density interventions across the three periods in the order of 80%, then 120%, then 100%.
- 100% Food Energy Density, Then 80%, Then 120%: Participants in the classroom that received the three food energy density interventions across the three periods in the order of 100%, then 80%, then 120%.
- 120% Food Energy Density, Then 100%, Then 80%: Participants in the classroom that received the three food energy density interventions across the three periods in the order of 120%, then 100%, then 80%.
Period: Study Week 1
Arm/Group | 80% Food Energy Density First, Then 100%, Then 120% | 100% Food Energy Density First, Then 120%, Then 80% | 120% Food Energy Density First, Then 80%, Then 100% | 80% Food Energy Density First, Then 120%, Then 100% | 100% Food Energy Density, Then 80%, Then 120% | 120% Food Energy Density, Then 100%, Then 80%
Started | 9 | 15 | 7 | 7 | 7 | 11
Completed | 7 | 14 | 7 | 5 | 7 | 11
Not Completed | 2 | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 2 | 0 | 0
Period: Study Week 2
Arm/Group | 80% Food Energy Density First, Then 100%, Then 120% | 100% Food Energy Density First, Then 120%, Then 80% | 120% Food Energy Density First, Then 80%, Then 100% | 80% Food Energy Density First, Then 120%, Then 100% | 100% Food Energy Density, Then 80%, Then 120% | 120% Food Energy Density, Then 100%, Then 80%
Started | 7 | 14 | 7 | 5 | 7 | 11
Completed | 7 | 14 | 7 | 5 | 7 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Study Week 3
Arm/Group | 80% Food Energy Density First, Then 100%, Then 120% | 100% Food Energy Density First, Then 120%, Then 80% | 120% Food Energy Density First, Then 80%, Then 100% | 80% Food Energy Density First, Then 120%, Then 100% | 100% Food Energy Density, Then 80%, Then 120% | 120% Food Energy Density, Then 100%, Then 80%
Started | 7 | 14 | 7 | 5 | 7 | 11
Completed | 7 | 14 | 7 | 4 | 7 | 11
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data of one participant was excluded from analysis due to absence from meals on three or more days of each 5-day study period.
Groups:
- All Study Participants: Enrolled participants who completed the trial and whose data was not excluded from analysis
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 5
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Differences in Food and Beverage Intake by Energy
Description: Differences in daily intake of food and beverages by energy, in kcal
Time Frame: Days 1-5 in Weeks 1, 2, and 3
Population: Data of 1 enrolled participant was excluded from analysis for absence from meals on 3 or more days in multiple intervention periods.
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | 100% Food Energy Density | 80% Food Energy Density | 120% Food Energy Density
Number analyzed (Participants) | 49 | 49 | 49
kilocalories | 956 (37) | 884 (38) | 1041 (38)
Statistical Analysis 1: Comparison: 100% Food Energy Density vs 80% Food Energy Density vs 120% Food Energy Density; Test type: Superiority; p < 0.0001, Mixed Models Analysis — According to predefined comparisons, outcomes of the 80% and 120% Food Energy Density interventions were compared to the outcome of the baseline (100%) intervention

2. Primary Outcome: Differences in Food and Beverage Intake by Weight
Description: Differences in daily intake of food and beverages by weight, in grams
Time Frame: Days 1-5 in weeks 1, 2, and 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: grams
Arm/Group | 100% Food Energy Density | 80% Food Energy Density | 120% Food Energy Density
Number analyzed (Participants) | 49 | 49 | 49
grams | 997 (41) | 952 (41) | 988 (41)
Statistical Analysis 1: Comparison: 100% Food Energy Density vs 80% Food Energy Density; Test type: Superiority; p = 0.10, Mixed Models Analysis — According to predefined comparisons, intake by weight in the 80% intervention was compared to the 100% intervention
Statistical Analysis 2: Comparison: 100% Food Energy Density vs 120% Food Energy Density; Test type: Superiority; p = 0.15, Mixed Models Analysis — According to predefined comparisons, intake by weight in the 120% intervention was compared to the 100% intervention

3. Secondary Outcome: Differences in Food and Beverage Intake by Energy Density
Description: Differences in daily intake of food and beverages by energy density, in kcal/g
Time Frame: Days 1-5 in weeks 1, 2, and 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilocalories/gram
Arm/Group | 100% Food Energy Density | 80% Food Energy Density | 120% Food Energy Density
Number analyzed (Participants) | 49 | 49 | 49
kilocalories/gram | 0.97 (0.02) | 0.93 (0.02) | 1.06 (0.03)
Statistical Analysis 1: Comparison: 100% Food Energy Density vs 80% Food Energy Density vs 120% Food Energy Density; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- 80% Food Energy Density: All participants during the 80% Food Energy Density intervention
- 100% Food Energy Density: All participants during the 100% Food Energy Density intervention
- 120% Food Energy Density: All participants during the 120% Food Energy Density intervention
Arm/Group | 80% Food Energy Density | 100% Food Energy Density | 120% Food Energy Density
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT03010501/Prot_SAP_000.pdf